CLINICAL TRIAL: NCT02881125
Title: A Phase 1 Study of Weekly Paclitaxel and Nortriptyline for Relapsed Small Cell Carcinoma
Brief Title: Paclitaxel and Nortriptyline Hydrochloride in Treating Patients With Relapsed Small Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9618; NCI-2016-01197 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9618 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Small Cell | interventions — Nortriptyline; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (paclitaxel, nortriptyline hydrochloride) (Experimental): Patients receive paclitaxel IV on days 1, 8, and 15. Patients also receive nortriptyline hydrochloride PO QD on days 1-7, BID on days 8-14, and TID on days 15-28 of course 1 and TID on days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nortriptyline Hydrochloride; Drug: Paclitaxel

INTERVENTIONS:
Drug: Nortriptyline Hydrochloride — Given PO
  Other Names: Allegron; Norpress; Pamelor
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase I trial studies the side effects and best dose of nortriptyline hydrochloride when given together with paclitaxel in treating patients with small cell carcinoma that has come back. Nortriptyline hydrochloride, may help disrupt survival signals and cause cancer cell death. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nortriptyline hydrochloride and paclitaxel may work better in treating patients with small cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) of nortriptyline hydrochloride (nortriptyline) combined with weekly paclitaxel (PC).

SECONDARY OBJECTIVES:

I. To assess the overall response rate (ORR) to nortriptyline combined with PC.

II. To assess progression free survival (PFS) and overall survival (OS).

OUTLINE: This is a dose-escalation study of nortriptyline hydrochloride.

Patients receive paclitaxel intravenously (IV) on days 1, 8, and 15. Patients also receive nortriptyline hydrochloride orally (PO) once daily (QD) on days 1-7, twice daily (BID) on days 8-14, and thrice daily (TID) on days 15-28 of course 1 and TID on days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days and every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent
* Pathologically-confirmed small cell carcinoma of any primary site
* Relapse following platinum-based chemotherapy or documented progressive disease while on platinum-based chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 at time of informed consent
* Absolute neutrophil count >= 1.5 x 10^9 cells/L
* Hemoglobin (Hgb) >= 9.0 g/dL
* Platelets >= 100,000 x 10^9/L
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Alkaline phosphatase levels =< 2.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN
* Serum creatinine < 1.5 mg/dL
* At least one site of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria on computed tomography (CT) scan done within 30 days prior to study start
* Women of child-bearing potential and sexually active men must agree to use adequate contraception (hormonal, barrier method, or abstinence) prior to study entry, during treatment, and for three months after completing treatment
* Baseline electrocardiogram demonstrating all of the following: corrected QT (QTc) < 450 milliseconds (msec) (men) and < 470 msec (women), PR < 240 msec, QRS < 100 msec

Exclusion Criteria:

* Untreated active major depression
* Bipolar disorder
* Pregnancy and lactation; refusal to use adequate contraception
* History of seizures in the past 3 years
* Concurrent therapy with monoamine oxidase inhibitors (MAOI), selective serotonin reuptake inhibitors (SSRI), or other tricyclic antidepressants (TCA) or use within 2 weeks study start
* Concomitant therapy with any drugs shown to have major interactions with nortriptyline (i.e. known inhibitors of cytochrome P450 family 2 subfamily D member 6 [CYP2D6]) and use during the 30-day period prior to study start
* Myocardial infarction in preceding 4 weeks; history of uncontrolled cardiac arrhythmias or family history of sudden cardiac death
* Peripheral neuropathy grade 2 or greater
* Progressive or symptomatic central nervous system (CNS) metastases; patients with known brain metastasis must have stable disease following treatment surgery, radiation, or both
* Glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose, determined by the number of patients who experience a dose limiting toxicity | Up to 28 days
  Maximum tolerated dose defined as the highest dose level of nortriptyline (in combination with weekly paclitaxel) where < 1/3 or < 2/6 patients experience a dose-limiting toxicity evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.

SECONDARY OUTCOMES:
Objective tumor response evaluated according to Response Evaluation Criteria in Solid Tumors version 1.1 | Up to 2 years
  Objective tumor response will be assessed with a 95% confidence interval.
Overall Survival | Up to 2 years
  Overall Survival will be described using Kaplan-Meier curves.
Progression free survival | Up to 2 years
  Progression free survival will be described using Kaplan-Meier curves.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montgomery, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States